CLINICAL TRIAL: NCT07088692
Title: Clinical Observation and Risk Factor Analysis of the Incidence of Postoperative PTSD in Children
Status: Not yet recruiting | Type: Observational
Sponsor: JianHao Zhang (Other)
Collaborators: Beijing Children's Hospital (Other); Capital Institute of Pediatrics, China (Other)
Responsible Party: Sponsor-Investigator, JianHao Zhang, postgraduate student, The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Organization: The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College (Other)
Other Study IDs: YS2024CG022
Record Dates: First submitted 2025-07-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: PTSD
Keywords: PTSD; PMTS
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Those who developed PTSD during the follow-up period after enrollment were categorized in the exposu: Those who did not develop PTSD during the follow-up period after enrollment were categorized as control group

SUMMARY:
Preoperative anxiety, pain, and repeated exposure to general anesthesia may increase the risk of post-traumatic stress disorder (PTSD) in children. This study aims to establish a clinical database by collecting the incidence and risk factors of PTSD in children aged 6 to 12 undergoing elective surgery under general anesthesia, with a primary focus on evaluating the overall postoperative PTSD incidence, its incidence at different time points, and identifying potential risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12 years scheduled for elective surgery under general anesthesia.
* Parent or legal guardian provides informed consent and agrees to complete a 1-year follow-up.

Exclusion Criteria:

* History of psychiatric disorders (e.g., PTSD, anxiety disorders), substance abuse, long-term use of steroids or hormonal medications.
* Significant cognitive impairment that hinders understanding of study procedures.
* Emergency surgery or trauma-related procedures requiring urgent general anesthesia.
* Recent (within two weeks) upper respiratory tract infection or severe pulmonary disease.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will enroll children aged 6 to 12 years scheduled for elective surgery under general anesthesia. Exclusion criteria include: a history of psychiatric disorders or significant cognitive impairment, recent upper respiratory tract infection or severe pulmonary disease (within the past two weeks), undergoing emergency surgery or trauma-related surgery under general anesthesia, or preoperative chronic pain.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Overall incidence of PTSD at different time points | 6 months
  Morbidity of enrolled children during follow-up assessed by CPSS questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- The Plastic Surgery Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-21): https://cdn.clinicaltrials.gov/large-docs/92/NCT07088692/Prot_SAP_000.pdf